CLINICAL TRIAL: NCT03097406
Title: Functional Outcome and Complications After Global Unite ® Prostheses in Osteoarthritis and Displaced Fractures of the Proximal Humerus.
Brief Title: Functional Outcome and Complications After Global Unite ® Prostheses
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Herlev and Gentofte Hospital (Other)
Collaborators: Zealand University Hospital (Other); DePuy Synthes (Industry)
Responsible Party: Principal Investigator, Alexander Amundsen, Principal investigator, Herlev and Gentofte Hospital
Other Study IDs: HERKOG2017
Record Dates: First submitted 2017-03-15; First posted 2017-03-31 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Osteoarthritis of the Shoulder; Proximal Humeral Fracture
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Osteoarthritis group: Patients with osteoarthritis (2017-2019) at Herlev Hospital treated with Global Unite total shoulder arthroplasty
  Interventions: Procedure: Global Unite total shoulder arthroplasty
- Osteoarthritis control group: Patients with osteoarthritis (2013-2016) at Herlev Hospital treated with a Global Advantage
  Interventions: Procedure: Global Advantage
- Fracture group: Patients with a fracture of the proximal humerus (2017-2019) at Køge and Herlev Hospital treated with Global Unite hemiarthroplasty
  Interventions: Procedure: Global Unite hemiarthroplasty
- Fracture control group: Patients with a fracture of the proximal humerus (2013-2016) at Køge and Herlev Hospital treated with Global FX hemiarthroplasty
  Interventions: Procedure: Global FX

INTERVENTIONS:
Procedure: Global Unite hemiarthroplasty — A hemiarthroplasty used for complex fractures of the proximal humerus.
  Groups: Fracture group
Procedure: Global Advantage — A total shoulder prosthesis used for osteoarthritis
  Groups: Osteoarthritis control group
Procedure: Global FX — A hemiarthroplasty used for complex fractures of the proximal humerus.
  Groups: Fracture control group
Procedure: Global Unite total shoulder arthroplasty — A total shoulder prosthesis used for osteoarthritis
  Groups: Osteoarthritis group

SUMMARY:
This study aims to investigate the shoulder function of patients with osteoarthritis or a fracture of the upper extremity after surgery with the Global Unite shoulder system.

The majority of fractures of the humerus are non-surgically treated, but for the complex cases where the fracture is irreparable (1), the treatment choice is a shoulder prosthesis called a hemiarthroplasty. Hemiarthroplasty has been associated to less pain and more quality of life , (2,3) but no difference in range of motion is reported when compared to non-surgically treatment of complex humeral fractures. (2,3,4)

One of the important steps in surgery of a fractured humerus is the fixation of the bone fragments in an anatomically correct position as previous studies have shown that complications related to the fixation and healing of bone fragments occurred in 11 % of patients treated with a hemiarthroplasty . The Global Unite hemiarthroplasty introduces a new feature, which allows the surgeon to more closely attach the bone fragments.

Patients with osteoarthritis and fractures of the humerus will be included from two hospitals, Herlev and Køge University Hospital. A total of 88 patients, 44 osteoarthritis and 44 fracture patients, are included. The patients will be followed two years after surgery and will be seen a total of four times postoperatively, where the function of the shoulder will be examined by questionnaires concerning shoulder function and quality of life, by a motion examination and by x-ray. The outcome of these examinations will be compared to the functional outcome of patients that have received different shoulder prostheses for the same diagnoses at Herlev and Køge University Hospital. The patients will undergo two radiographic scans after surgery, to determine whether or not bone fragments remain in an anatomically correct position in the patients with a fracture of the proximal humerus. A special focus will be on the function of the shoulder in patients with bone fragments that are not in an anatomically correct position. Furthermore, complications and the need of reoperation were registered during the two-year follow-up period.

The aims of this study is to

* Determine the function of the shoulder in patients receiving the Global Unite prosthesis due to either osteoarthritis or fracture of the humerus.
* To compare these results with results from patients previously treated with a different prosthesis designs
* To determine the influence of the fixation of bone fragments in the postoperative function in fracture patients.

DETAILED DESCRIPTION:
The study was based on data from Køge and Herlev University Hospital. All patients that fit the inclusion criteria and had an indication for shoulder replacement where included and the study started on the 1st of January 2017.

Aim

* To determine 2-year postoperative outcome, complications and revision rates in patients receiving a Global Unite
* To compare the postoperative outcome to patients from a in matched control group
* To determine the influence of tuberosity placement and migration on functional outcome in patients with a fracture of the proximal humerus.

The trauma mechanism of the fractures and health status of the patients were determined upon arrival. A preoperative CT-scan was performed in all fracture patients for preoperative planning. A CT-scan was also performed preoperatively in the osteoarthritis patients to determine the degree of bone degeneration. An x-ray was performed right after surgery, 3 months and 24 months postoperatively.

The patients included received a Global Unite hemiarthroplasty in the fracture situation and a Global Unite total shoulder in osteoarthritis patients. The patients received standardized postoperative analgesic treatment and physiotherapy rehabilitation and all patients had postoperative follow-up 3, 6 months, 1-year and 2-year after surgery. The outcome at the follow-up was determined by using Oxford Shoulder Score, Constant-Murley score, EQ-5-D questionnaire and Western Ontario Osteoarthritis of the Shoulder index

Factors like American Society of Anesthesiologists score, body-mass index, smoking, alcohol, medication and comorbidity were registered. Furthermore time from injury to surgery, surgery time, length of hospital stay, complications (osteonecrosis, infection, loosening), revision, discharge type, pain score and analgesia were reported. The preoperatively function was only registered for osteoarthritis patients.

The study was performed as a prospective cohort study with a historic control group. The fracture patients submitted for a Global Unite from February 2017 were compared to fracture patients receiving the Global FX at Herlev and Køge Hospital from 2013 to 2016 and the osteoarthritis patients receiving a Global Unite total shoulder were compared to patients receiving a Global Advantage at Herlev Hospital from 2013-2016. 44 patients were included in the control and the intervention groups, of both diagnoses, to obtain power of 80 % in power calculations based on Constant-Murley score. This equals a total of 88 patients in the intervention groups and 88 patients in the control groups. It was estimated that it would take 2 to 3 years to include osteoarthritis- and fracture-patients in this study.

All surgery was performed by 5 senior consultants at Herlev Hospital and 2 senior consultants at Køge Hospital. The postoperative functional outcome of patients in the first half of the study was compared to the outcome of patients in the last half to determine a possible learning curve. The follow-up was performed by one independent physician

ELIGIBILITY:
Inclusion Criteria:

Osteoarthritis patients:

* Pronounced osteoarthritis
* physician-assessed need of surgery
* Surgery at Herlev University Hospital

Fracture patients:

* Luxation fractures
* 4-part fractures
* Displaced 3-part fractures
* Headsplit fractures
* Treated at Herlev University Hospital or Køge University Hospital

Control group:

* Surgery from 2013-2017
* Treated for osteoarthritis with Global Advantage
* Osteoarthritis surgery at Herlev University Hospital
* Treated with Global FX due to fracture of the proximal humerus
* Global FX treatment at Herlev or Køge University Hospital

Exclusion Criteria:

* Patients not living in Denmark
* Two-part fractures of the proximal humerus
* Patient without a Danish civil registration number
* Patients younger than 50
* Revision surgery
* Previous arthroplasty procedures in the same shoulder
* Deceased patients

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The fracture patients will be included from the emergency rooms and outpatient visits at Herlev and Køge University Hospital. Patients are assessed by experienced shoulder surgeons before surgery.
  Osteoarthritis patients are assessed by outpatient visits to Herlev University Hospital.
  The fracture and osteoarthritis control groups are found in the hospitals' registries and are offered an inspection of the shoulder.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Functional outcome (Western Ontario Osteoarthritis of the Shoulder (WOOS)) | 3 months after surgery
  The WOOS questionnaire is used to measure the patient-reported functional outcome for the patients.
Functional outcome (Western Ontario Osteoarthritis of the Shoulder (WOOS)) | 6 months after surgery
  The WOOS questionnaire is used to measure the patient-reported functional outcome for the patients.
Functional outcome (Western Ontario Osteoarthritis of the Shoulder (WOOS)) | 12 months after surgery
  The WOOS questionnaire is used to measure the patient-reported functional outcome for the patients. . The outcome will be compared with outcome of patients that previously received Global FX or Global Advantage for fracture or osteoarthritis, respectively.
Functional outcome (Western Ontario Osteoarthritis of the Shoulder (WOOS)) | 24 months after surgery
  The WOOS questionnaire is used to measure the patient-reported functional outcome for the patients. The outcome will be compared with outcome of patients that previously received Global FX or Global Advantage for fracture or osteoarthritis, respectively.
Functional outcome (Constant-Murley Score (CMS)) | 3 months after surgery
  CMS is used to measure the functional outcome for the patients.
Functional outcome (Constant-Murley Score (CMS)) | 6 months after surgery
  CMS is used to measure the functional outcome for the patients.
Functional outcome (Constant-Murley Score (CMS)) | 12 months after surgery
  CMS is used to measure the functional outcome for the patients.
Functional outcome (Constant-Murley Score (CMS)) | 24 months after surgery
  CMS is used to measure the functional outcome for the patients. The outcome will be compared with outcome of patients that previously received Global FX or Global Advantage for fracture or osteoarthritis, respectively
Functional outcome (Oxford Shoulder Score (OSS)) | 3 months after surgery
  The OSS questionnaire is used to measure the patient-reported functional outcome.
Functional outcome (Oxford Shoulder Score (OSS)) | 6 months after surgery
  The OSS questionnaire is used to measure the patient-reported functional outcome.
Functional outcome (Oxford Shoulder Score (OSS)) | 12 months after surgery
  The OSS questionnaire is used to measure the patient-reported functional outcome.
Functional outcome (Oxford Shoulder Score (OSS)) | 24 months after surgery
  The OSS questionnaire is used to measure the patient-reported functional outcome. The outcome will be compared with outcome of patients that previously received Global FX or Global Advantage for fracture or osteoarthritis, respectively

SECONDARY OUTCOMES:
Tuberosity migration or vanishing in fracture patients | Baseline CT-scan, x-rays 3 and 24 months after surgery
  A preoperative CT-scan will be performed and postoperative x-rays will be performed to determine whether or not the tuberosities have migrated or vanished in the fracture patients treated with Global Unite hemiarthroplasty

OTHER OUTCOMES:
Complications | Up to 24 months after surgery, the last record is made in December 2021
  Complications(infections, loosening etc) will be registered during this prospective study.
Revisions | Up to 24 months after surgery, the last record is made in December 2021
  Patients who undergo revision surgery are registered and the revision rate will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Amundsen, MD, Principal Investigator — University of Copenhagen
Locations (2):
- Denmark (2):
  - Herlev University Hospital, Herlev, Copenhagen
  - Køge University Hospital, Køge

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bryant D, Litchfield R, Sandow M, Gartsman GM, Guyatt G, Kirkley A. A comparison of pain, strength, range of motion, and functional outcomes after hemiarthroplasty and total shoulder arthroplasty in patients with osteoarthritis of the shoulder. A systematic review and meta-analysis. J Bone Joint Surg Am. 2005 Sep;87(9):1947-56. doi: 10.2106/JBJS.D.02854. PMID 16140808
- [Background] Olerud P, Ahrengart L, Ponzer S, Saving J, Tidermark J. Hemiarthroplasty versus nonoperative treatment of displaced 4-part proximal humeral fractures in elderly patients: a randomized controlled trial. J Shoulder Elbow Surg. 2011 Oct;20(7):1025-33. doi: 10.1016/j.jse.2011.04.016. Epub 2011 Jul 23. PMID 21783385
- [Background] den Hartog D, de Haan J, Schep NW, Tuinebreijer WE. Primary shoulder arthroplasty versus conservative treatment for comminuted proximal humeral fractures: a systematic literature review. Open Orthop J. 2010 Feb 17;4:87-92. doi: 10.2174/1874325001004020087. PMID 20309406
- [Background] Handoll HH, Ollivere BJ, Rollins KE. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2012 Dec 12;12:CD000434. doi: 10.1002/14651858.CD000434.pub3. PMID 23235575